CLINICAL TRIAL: NCT00094107
Title: Phase 2 Study Of The Anti-Angiogenesis Agent AG-013736 In Patients With Metastatic Melanoma
Brief Title: Anti-Angiogenesis Agent AG-013736 In Patients With Metastatic Melanoma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: A4061015
Record Dates: First submitted 2004-10-11; First posted 2004-10-14 (Estimated); Results first posted 2012-03-30 (Estimated); Last update posted 2012-06-26 (Estimated); Status verified 2012-06

CONDITIONS: Melanoma; Skin Neoplasms
Keywords: melanoma; antiangiogenesis
MeSH Terms: conditions — Melanoma; Skin Neoplasms | interventions — Axitinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Axitinib [AG-013736] (Experimental)
  Interventions: Drug: Axitinib [AG-013736]

INTERVENTIONS:
Drug: Axitinib [AG-013736] — VEGFR [vascular endothelial growth factor Receptor] and PDGFR [Platelet-Derived Growth Factor Receptor] inhibitor: Single agent AG-013736 starting dose 5 mg BID +/- 20% according to toxicity. Treatment until progression or unacceptable toxicity occurs.

SUMMARY:
This is a Phase 2 study being conducted at multiple centers in the United States and France. Patients having melanoma that has spread to other parts of the body (i.e., metastatic) are eligible to participate. Patients must have disease that has been treated with no more than 1 prior treatment for metastatic disease (prior adjuvant treatment for localized disease does not count as prior treatment for metastatic disease). The purpose of the study is to test whether the angiogenesis inhibitor AG-013736 is an effective treatment for metastatic melanoma as shown by the number of patients in the study who experience significant and durable tumor shrinkage.

ELIGIBILITY:
Inclusion Criteria:

* Histologically documented melanoma with metastases
* No more than 1 prior systemic therapy for metastatic disease (prior adjuvant therapy with interferon does not count as prior therapy for metastatic disease)

Exclusion Criteria:

* History of hemoptysis (coughing up of blood)
* Brain metastases

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2004-12; Primary Completion 2008-04 (Actual); Study Completion 2008-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (9):
- United States (8):
  - Pfizer Investigational Site, Orange, California
  - Pfizer Investigational Site, Miami Beach, Florida
  - Pfizer Investigational Site, Boston, Massachusetts
  - Pfizer Investigational Site, Clairton, Pennsylvania
  - Pfizer Investigational Site, Greensburg, Pennsylvania
  - Pfizer Investigational Site, Johnstown, Pennsylvania
  - Pfizer Investigational Site, Pittsburgh, Pennsylvania
  - Pfizer Investigational Site, Wexford, Pennsylvania
- Pfizer Investigational Site, Paris, France

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=A4061015&StudyName=Anti-Angiogenesis%20Agent%20AG-013736%20In%20Patients%20With%20Metastatic%20Melanoma

RESULTS

PARTICIPANT FLOW:
Groups:
- Axitinib: Axitinib (AG-013736) tablet administered orally at a dose of 5 milligram (mg) twice daily (BID) in cycles of 4 weeks. Treatment was administered continuously until progression or unacceptable toxicity occurred.
Period: Overall Study
Arm/Group | Axitinib
Started | 32
Completed | 0
Not Completed | 32
Not completed — Lack of Efficacy | 23
Not completed — Death | 5
Not completed — Adverse Event | 3
Not completed — Withdrawal due to Disease Progression | 1

BASELINE CHARACTERISTICS:
Groups:
- Axitinib: Axitinib (AG-013736) tablet administered orally at a dose of 5 mg BID in cycles of 4 weeks. Treatment was administered continuously until progression or unacceptable toxicity occurred.
Arm/Group | Axitinib
Number analyzed (Participants) | 32
Age Continuous [Mean (Standard Deviation); unit: Years] | 62.40 (15.56)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 15
  Male | 17

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Objective Response (OR)
Description: Percentage of participants with OR based assessment of confirmed complete response (CR) or confirmed partial response (PR) according to Response Evaluation Criteria in Solid Tumors (RECIST). Confirmed responses are those that persist on repeat imaging study at least 4 weeks after initial documentation of response. CR are defined as the disappearance of all lesions (target and/or non target). PR are those with at least 30 percent (%) decrease in the sum of the longest dimensions of the target lesions taking as a reference the baseline sum longest dimensions.
Time Frame: Baseline until the date of first documented progression or discontinuation from the study due to any cause, assessed every 8 weeks up to 147 weeks
Population: Study population included all participants who received at least 1 dose of study medication and had at least one baseline efficacy assessment.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Axitinib
Number analyzed (Participants) | 32
Percentage of participants | 18.8 [7.2 to 36.4]

2. Secondary Outcome: Progression-free Survival (PFS)
Description: Time in days from start of study treatment to first documentation of objective tumor progression or death due to any cause. PFS was calculated as first event date minus the date of first dose of study medication plus 1. Tumor progression was determined from oncologic assessment data (where data meet the criteria for progressive disease [PD]), or from adverse event (AE) data (where the outcome was "Death").
Time Frame: Baseline until the date of first documented progression or death due to any cause, assessed every 8 weeks up to 147 weeks
Population: as for outcome 1
Measure: Median (95% Confidence Interval); unit: Days
Arm/Group | Axitinib
Number analyzed (Participants) | 32
Days | 117.5 [69.0 to 204.0]

3. Secondary Outcome: Duration of Response (DR)
Description: Time in days from the first documentation of objective tumor response to objective tumor progression or death due to any cause. Duration of tumor response was calculated as the date of the first documentation of objective tumor progression or death due to cancer minus the date of the first CR or PR that was subsequently confirmed plus 1. DR was calculated for the subgroup of participants with a confirmed objective tumor response.
Time Frame: as for outcome 1
Population: Subgroup of participants from the study population with a confirmed objective tumor response (CR or PR).
Measure: Median (95% Confidence Interval); unit: Days
Arm/Group | Axitinib
Number analyzed (Participants) | 5
Days | 179.0 [151.0 to 516.0]

4. Secondary Outcome: Overall Survival (OS)
Description: Time in days from the start of study treatment to date of death due to any cause. OS was calculated as the death date minus the date of first dose of study medication plus 1. Death was determined from AE data (where outcome was death) or from follow-up contact data (where the participant current status was death). For participants who were alive, overall survival was censored at the last contact.
Time Frame: Baseline to death due to any cause or at least 1 year after the initial dose for the last treated participant
Population: Study population included all participants who received at least 1 dose of study medication.
Measure: Median (95% Confidence Interval); unit: Days
Arm/Group | Axitinib
Number analyzed (Participants) | 32
Days | 200.5 [157.0 to 274.0]

5. Other Pre Specified Outcome: Population Pharmacokinetics for Axitinib (AG-013736) Plasma Concentrations
Description: Population pharmacokinetic analysis involved mixed effects modeling using nonlinear mixed effects modeling (NONMEM) software. The intent of this analysis was to establish a basic population pharmacokinetic model for axitinib (AG-013736) and to determine inter-individual and residual variability in population (oral) clearance, and volume of distribution of drug. Relationship of demographic variables (gender, age, body weight, height and ethnicity), concomitant medications and measures of altered hepatic and renal function were examined by fitting measured axitinib (AG-013736) concentrations.
Time Frame: Day 1 (pre-dose), Day 29, Day 57 and then every 8 weeks up to 147 weeks
Population: Population pharmacokinetic values were not summarized as descriptive statistics since the data was not available for the single study and data for all the axitinib (AG-013736) Phase 2 studies would be pooled together in a separate report.
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Axitinib
Number analyzed (Participants) | 0

6. Other Pre Specified Outcome: Plasma Concentrations of Soluble Proteins
Description: Plasma concentrations of soluble proteins (vascular endothelial growth factor [VEGF], placental growth factor [PlGF] and soluble vascular endothelial growth factor receptor-2 [sVEGFR2]) may be associated with tumor angiogenesis or tumor physiology and may correlate with efficacy or biological activity. It is presented as ratio to baseline, which is obtained by dividing the plasma soluble protein concentration at each time point by its concentration at baseline.
Time Frame: Day 1 (pre-dose) and then every 8 weeks up to 147 weeks
Population: Ratio to baseline values for plasma soluble proteins were not summarized as descriptive statistics since the data was not available for the single study and data for all the axitinib Phase 2 studies would be pooled together in a separate report.
Measure: Mean (Standard Deviation); unit: Ratio
Arm/Group | Axitinib
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Description: The same event may appear as both an AE and a SAE. However, what is presented are distinct events. An event may be categorized as serious in one subject and as nonserious in another subject, or one subject may have experienced both a serious and nonserious event during the study.
Arm/Group | Axitinib
Serious Adverse Events (participants affected / at risk) | 18/32
Other Adverse Events (participants affected / at risk) | 32/32
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Axitinib (N=32)
Atrial fibrillation (Cardiac disorders) | 1
Atrial tachycardia (Cardiac disorders) | 1
Cardiac arrest (Cardiac disorders) | 1
Abdominal pain, not otherwise specified (NOS) (Gastrointestinal disorders) | 1
Intestinal perforation NOS (Gastrointestinal disorders) | 1
Disease progression NOS (General disorders) | 1
Fatigue (General disorders) | 1
General physical health deterioration (General disorders) | 2
Pain NOS (General disorders) | 1
Cholestasis (Hepatobiliary disorders) | 1
Aspergillosis (Infections and infestations) | 1
Pneumonia NOS (Infections and infestations) | 1
Sepsis NOS (Infections and infestations) | 1
Staphylococcal bacteraemia (Infections and infestations) | 1
Staphylococcal sepsis (Infections and infestations) | 1
Jaw fracture (Injury, poisoning and procedural complications) | 1
Blood lactate dehydrogenase increased (Investigations) | 1
Transaminases increased (Investigations) | 1
Anorexia (Metabolism and nutrition disorders) | 1
Dehydration (Metabolism and nutrition disorders) | 2
Diabetes mellitus inadequate control (Metabolism and nutrition disorders) | 1
Failure to thrive (Metabolism and nutrition disorders) | 1
Malignant pleural effusion (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Cerebrovascular accident (Nervous system disorders) | 1
Confusion (Psychiatric disorders) | 1
Depression (Psychiatric disorders) | 1
Renal artery stenosis (Renal and urinary disorders) | 1
Dyspnoea NOS (Respiratory, thoracic and mediastinal disorders) | 1
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 2
Respiratory arrest (Respiratory, thoracic and mediastinal disorders) | 1
Hypertension NOS (Vascular disorders) | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Axitinib (N=32)
Leukocytosis (Blood and lymphatic system disorders) | 1
Tachycardia (Cardiac disorders) | 1
Deafness (Ear and labyrinth disorders) | 1
Ear congestion (Ear and labyrinth disorders) | 1
Tinnitus (Ear and labyrinth disorders) | 1
Hypothyroidism (Endocrine disorders) | 3
Conjunctivitis (Eye disorders) | 1
Eyelid ptosis (Eye disorders) | 1
Visual impairment (Eye disorders) | 2
Abdominal discomfort (Gastrointestinal disorders) | 2
Abdominal distension (Gastrointestinal disorders) | 1
Abdominal pain (Gastrointestinal disorders) | 3
Abdominal pain upper (Gastrointestinal disorders) | 2
Abdominal tenderness (Gastrointestinal disorders) | 1
Anal inflammation (Gastrointestinal disorders) | 1
Constipation (Gastrointestinal disorders) | 7
Diarrhoea (Gastrointestinal disorders) | 11
Diverticulum intestinal (Gastrointestinal disorders) | 1
Dry mouth (Gastrointestinal disorders) | 3
Dyspepsia (Gastrointestinal disorders) | 4
Dysphagia (Gastrointestinal disorders) | 2
Flatulence (Gastrointestinal disorders) | 1
Gastritis (Gastrointestinal disorders) | 1
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 2
Intestinal perforation (Gastrointestinal disorders) | 1
Nausea (Gastrointestinal disorders) | 13
Odynophagia (Gastrointestinal disorders) | 1
Oesophagitis (Gastrointestinal disorders) | 1
Oral pain (Gastrointestinal disorders) | 2
Retching (Gastrointestinal disorders) | 1
Stomatitis (Gastrointestinal disorders) | 4
Vomiting (Gastrointestinal disorders) | 7
Asthenia (General disorders) | 10
Chest discomfort (General disorders) | 1
Fat tissue increased (General disorders) | 1
Fatigue (General disorders) | 20
Feeling hot (General disorders) | 1
General physical health deterioration (General disorders) | 2
Impaired healing (General disorders) | 1
Malaise (General disorders) | 3
Mucosal inflammation (General disorders) | 4
Oedema peripheral (General disorders) | 5
Pain (General disorders) | 2
Pyrexia (General disorders) | 4
Hepatic pain (Hepatobiliary disorders) | 2
Hepatomegaly (Hepatobiliary disorders) | 1
Drug hypersensitivity (Immune system disorders) | 1
Seasonal allergy (Immune system disorders) | 1
Bronchitis (Infections and infestations) | 1
Device related infection (Infections and infestations) | 1
Gastroenteritis (Infections and infestations) | 1
Nasopharyngitis (Infections and infestations) | 1
Rhinitis (Infections and infestations) | 1
Sinusitis (Infections and infestations) | 1
Upper respiratory tract infection (Infections and infestations) | 1
Urinary tract infection (Infections and infestations) | 7
Fall (Injury, poisoning and procedural complications) | 1
Post procedural haemorrhage (Injury, poisoning and procedural complications) | 1
Vascular graft complication (Injury, poisoning and procedural complications) | 1
Alanine aminotransferase increased (Investigations) | 1
Aspartate aminotransferase increased (Investigations) | 1
Blood bilirubin increased (Investigations) | 1
Blood lactate dehydrogenase increased (Investigations) | 1
Transaminases increased (Investigations) | 1
Urine output decreased (Investigations) | 1
Weight decreased (Investigations) | 8
Decreased appetite (Metabolism and nutrition disorders) | 11
Dehydration (Metabolism and nutrition disorders) | 4
Hypercalcaemia (Metabolism and nutrition disorders) | 1
Hypokalaemia (Metabolism and nutrition disorders) | 1
Hypomagnesaemia (Metabolism and nutrition disorders) | 1
Hypophagia (Metabolism and nutrition disorders) | 2
Arthralgia (Musculoskeletal and connective tissue disorders) | 7
Back pain (Musculoskeletal and connective tissue disorders) | 4
Bone disorder (Musculoskeletal and connective tissue disorders) | 1
Bone pain (Musculoskeletal and connective tissue disorders) | 1
Flank pain (Musculoskeletal and connective tissue disorders) | 1
Groin pain (Musculoskeletal and connective tissue disorders) | 2
Muscular weakness (Musculoskeletal and connective tissue disorders) | 3
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 2
Musculoskeletal discomfort (Musculoskeletal and connective tissue disorders) | 2
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 2
Musculoskeletal stiffness (Musculoskeletal and connective tissue disorders) | 1
Myalgia (Musculoskeletal and connective tissue disorders) | 3
Neck pain (Musculoskeletal and connective tissue disorders) | 1
Nodule on extremity (Musculoskeletal and connective tissue disorders) | 1
Pain in extremity (Musculoskeletal and connective tissue disorders) | 8
Pain in jaw (Musculoskeletal and connective tissue disorders) | 1
Sensation of heaviness (Musculoskeletal and connective tissue disorders) | 1
Tendonitis (Musculoskeletal and connective tissue disorders) | 1
Lung neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Metastatic pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Vulval neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Balance disorder (Nervous system disorders) | 1
Cognitive disorder (Nervous system disorders) | 1
Dizziness (Nervous system disorders) | 6
Dysarthria (Nervous system disorders) | 1
Dysgeusia (Nervous system disorders) | 5
Headache (Nervous system disorders) | 6
Hyperaesthesia (Nervous system disorders) | 1
Hypogeusia (Nervous system disorders) | 1
Memory impairment (Nervous system disorders) | 1
Mental impairment (Nervous system disorders) | 1
Paraesthesia (Nervous system disorders) | 4
Peripheral sensory neuropathy (Nervous system disorders) | 1
Somnolence (Nervous system disorders) | 1
Spinal cord compression (Nervous system disorders) | 1
Agitation (Psychiatric disorders) | 2
Anhedonia (Psychiatric disorders) | 1
Anxiety (Psychiatric disorders) | 3
Depression (Psychiatric disorders) | 7
Hallucination (Psychiatric disorders) | 1
Insomnia (Psychiatric disorders) | 8
Mental status changes (Psychiatric disorders) | 2
Mood altered (Psychiatric disorders) | 1
Pollakiuria (Renal and urinary disorders) | 1
Proteinuria (Renal and urinary disorders) | 2
Amenorrhoea (Reproductive system and breast disorders) | 1
Benign prostatic hyperplasia (Reproductive system and breast disorders) | 1
Breast mass (Reproductive system and breast disorders) | 1
Menopausal symptoms (Reproductive system and breast disorders) | 1
Oedema genital (Reproductive system and breast disorders) | 1
Scrotal oedema (Reproductive system and breast disorders) | 1
Vaginal haemorrhage (Reproductive system and breast disorders) | 2
Cough (Respiratory, thoracic and mediastinal disorders) | 6
Dry throat (Respiratory, thoracic and mediastinal disorders) | 1
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 12
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 6
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 2
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 2
Hiccups (Respiratory, thoracic and mediastinal disorders) | 1
Hyperventilation (Respiratory, thoracic and mediastinal disorders) | 1
Lung disorder (Respiratory, thoracic and mediastinal disorders) | 1
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1
Pleuritic pain (Respiratory, thoracic and mediastinal disorders) | 2
Productive cough (Respiratory, thoracic and mediastinal disorders) | 1
Alopecia (Skin and subcutaneous tissue disorders) | 3
Blister (Skin and subcutaneous tissue disorders) | 2
Decubitus ulcer (Skin and subcutaneous tissue disorders) | 1
Dermatitis contact (Skin and subcutaneous tissue disorders) | 1
Dry skin (Skin and subcutaneous tissue disorders) | 2
Erythema (Skin and subcutaneous tissue disorders) | 3
Exfoliative rash (Skin and subcutaneous tissue disorders) | 1
Nail disorder (Skin and subcutaneous tissue disorders) | 2
Night sweats (Skin and subcutaneous tissue disorders) | 1
Pain of skin (Skin and subcutaneous tissue disorders) | 1
Palmar-plantar erythrodysaesthesia syndrome (Skin and subcutaneous tissue disorders) | 5
Plantar erythema (Skin and subcutaneous tissue disorders) | 1
Pruritus (Skin and subcutaneous tissue disorders) | 1
Rash (Skin and subcutaneous tissue disorders) | 3
Skin discomfort (Skin and subcutaneous tissue disorders) | 1
Skin lesion (Skin and subcutaneous tissue disorders) | 1
Skin warm (Skin and subcutaneous tissue disorders) | 1
Urticaria (Skin and subcutaneous tissue disorders) | 1
Menopause (Social circumstances) | 1
Skin neoplasm excision (Surgical and medical procedures) | 2
Haematoma (Vascular disorders) | 1
Hot flush (Vascular disorders) | 2
Hypertension (Vascular disorders) | 14
Iliac artery stenosis (Vascular disorders) | 1
Orthostatic hypotension (Vascular disorders) | 1

LIMITATIONS AND CAVEATS:
Population pharmacokinetic and plasma concentrations of soluble proteins were not presented, as the data was not available for the single study and data for all the axitinib (AG-013736) Phase 2 studies would be pooled together in a separate report.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), less than 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.